CLINICAL TRIAL: NCT06775665
Title: Clinical Characteristics and Real-World Outcomes of Chinese Patients With Hypertrophic Cardiomyopathy: A Prospective Cohort Study
Brief Title: A Real-World Study on Hypertrophic Cardiomyopathy in Chinese Population
Acronym: HCM
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-1249
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-01

CONDITIONS: Hypertrophic Cardiomyopathy (HCM)
Keywords: hypertrophic cardiomyopathy; real-world study
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HCM: Patients diagnosed with hypertrophic cardiomyopathy (HCM) according to the 2023 Guideline for Diagnosis and Treatment of Patients With Hypertrophic Cardiomyopathy were consecutively enrolled. These patients received pharmacological, interventional, or surgical treatment based on real-world treatment strategies. Follow-up was conducted to observe patient prognosis and the occurrence of outcome events.
  Interventions: Other: No interventions were applied to the patients.

INTERVENTIONS:
Other: No interventions were applied to the patients. — No interventions were applied to the patients.

SUMMARY:
This study is a prospective cohort study aimed at exploring the baseline characteristics and treatment patterns of the Chinese population with hypertrophic cardiomyopathy (HCM) in real-world settings. The objective is to assess the real-world treatment approaches and longitudinal outcomes in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent (ICF) and any required privacy authorization before the start of the study.
2. Aged ≥18 years at the time of signing the written informed consent.
3. Diagnosed with hypertrophic cardiomyopathy (HCM) according to the 2023 Guideline for Diagnosis and Treatment of Patients With Hypertrophic Cardiomyopathy, meeting the following criteria:

   1. Left ventricular wall thickness ≥15 mm in any segment at end-diastole, as assessed by echocardiography or cardiac magnetic resonance imaging (MRI).
   2. Left ventricular wall thickness ≥13 mm in individuals with a positive pathogenic gene test or those identified as members of a genetically affected family.
   3. Exclusion of other cardiovascular diseases or systemic/metabolic diseases causing ventricular wall thickening.

Exclusion Criteria:

1. Uncontrolled primary hypertension.
2. Moderate or severe aortic valve stenosis and/or primary mitral valve disease with severe mitral regurgitation.
3. Confirmed infiltrative or storage diseases with a phenotype resembling hypertrophic cardiomyopathy (e.g., Fabry disease, amyloidosis).
4. Expected life expectancy <1 years.
5. Severe infections, liver failure, renal failure, or other life-threatening conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hypertrophic cardiomyopathy
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2031-01-01 (Estimated); Study Completion 2032-06-01 (Estimated)

PRIMARY OUTCOMES:
Composite Cardiovascular Endpoints | 5 years
  Number of Participants with a composite cardiovascular endpoint consisting of ischemic stroke, heart failure hospitalization, and cardiovascular death

SECONDARY OUTCOMES:
All-cause mortality | 5 years
  Rate of death resulting from any cause, encompassing both disease-related and non-disease-related factors
Cardiovascular death | 5 years
  Rate of death resulting from cardiac diseases
New-onset arrhythmia | 5 years
  Number of Participants with new-onset arrhythmia
Sudden cardiac death (SCD) | 5 years
  Number of Participants suffer from sudden cardiac death
Non-fatal acute myocardial infarction | 5 years
  Number of Participants suffer from non-fatal acute myocardial infarction
Ischemic stroke | 5 years
  Number of participants suffer from ischemic stroke
Heart failure hospitalization | 5 years
  The rehospitalization rate of participants due to heart failure
New York Heart Association (NYHA) Classification | 5 years
  Percentage of participants with changes in NYHA classification
Kansas City Cardiomyopathy Questionnaire-23 (KCCQ-23) | 5 years
  The KCCQ-23 is a disease-specific health status assessment tool consisting of 23 items that quantify physical limitation, symptoms, self-efficacy, social limitation, and quality of life related to heart failure. Scores range from 0 to 100, with higher scores indicating better health status
BNP/NT-proBNP | 5 years
  Changes in serum BNP/NT-proBNP concentrations compared to baseline
Troponin T/I | 5 years
  Changes in serum cardiac troponin concentrations compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojie Xie, PhD, Principal Investigator — Second Affiliated Hospital, Zhejiang University School of Medicine
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided